CLINICAL TRIAL: NCT04502966
Title: Grass Pollen Sublingual Tablet Immunotherapy Plus Dupilumab for Induction of Tolerance in Adults With Moderate to Severe Seasonal Allergic Rhinitis (ITN084AD)
Brief Title: Grass Pollen Immunotherapy Plus Dupilumab for Tolerance Induction
Acronym: GRADUATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); ALK-Abelló A/S (Industry); Regeneron Pharmaceuticals (Industry); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ITN084AD; NIAID CRMS ID#: 38629 (Other: DAIT NIAID); 2018-003456-20 (EudraCT Number)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Allergic Rhinoconjunctivitis; Grass Pollen Allergy
Keywords: immunotherapy; nasal allergen challenge (NAC); total nasal symptom score (TNSS)
MeSH Terms: interventions — dupilumab; Grazax; Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grazax® +Dupixent® (Experimental): Participants randomized to this assignment will receive the following during the initial 2-year period of the trial:
  * Once daily tablet of Grazax® sublingual immunotherapy and
  * Dupixent® administered every other week (e.g., biweekly) by subcutaneous injection
  Interventions: Biological: Dupixent®; Biological: Grazax®
- Grazax® + Dupixent® Placebo (Experimental): Participants randomized to this assignment will receive the following during the initial 2-year period of the trial:
  * Once daily tablet of Grazax® sublingual immunotherapy and
  * Placebo for Dupixent® administered every other week (e.g., biweekly) by subcutaneous injection
  Interventions: Biological: Grazax®; Drug: Dupixent® Placebo
- Grazax® Placebo +Dupixent® Placebo (Placebo Comparator): Participants randomized to this assignment will receive the following during the initial 2-year period of the trial:
  * Once daily tablet of placebo for Grazax® sublingual immunotherapy and
  * Placebo for Dupixent® administered every other week (e.g., biweekly) by subcutaneous injection
  Interventions: Drug: Dupixent® Placebo; Drug: Grazax® Placebo

INTERVENTIONS:
Biological: Dupixent® — An initial dose of 600 mg (two 300 mg injections), followed by 300 mg administered every other week (biweekly), by subcutaneous injection.
  Other Names: dupilumab; monoclonal antibody against the IL-4 receptor
  Arms: Grazax® +Dupixent®
Biological: Grazax® — One Grazax® tablet daily, by sublingual administration.
  Grazax® is formulated as a freeze-dried oral lyophilisate/orally disintegrating tablet for oromucosal use. The active pharmaceutical ingredient is a standardized allergen extract derived from extraction and purification of grass pollen from timothy grass (Phleum pratense). The biological activity of the allergen is expressed in Standardized Quality Tablet units (SQ-T) units. The Grazax® dosage is one oral lyophilisate (75,000 Standardized Quality Tablet units (SQ-T) or approximately 2800 Bioequivalent allergy units (BAU), a measure of Phleum pratense SQ total biological potency defined by the FDA.
  Other Names: grass pollen allergen sublingual immunotherapy (SLIT); timothy grass (Phleum pratense) sublingual immunotherapy (SLIT)
  Arms: Grazax® + Dupixent® Placebo; Grazax® +Dupixent®
Drug: Dupixent® Placebo — Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose followed by a single injection administered every other week.
  Dupixent® placebo is a subcutaneous injection whose composition is identical to the active Dupixent®, with the exception of the active pharmaceutical ingredient.
  Other Names: placebo
  Arms: Grazax® + Dupixent® Placebo; Grazax® Placebo +Dupixent® Placebo
Drug: Grazax® Placebo — One tablet of Placebo (for Grazax®) daily, by sublingual administration.
  Grazax® placebo is a tablet whose composition is identical to the active Grazax® tablet with the only exception being exclusion of the active pharmaceutical ingredient, Phleum pratense Standardized Quality Tablet (SQ-T) units.
  Other Names: placebo
  Arms: Grazax® Placebo +Dupixent® Placebo

SUMMARY:
The primary objective of this study is to assess whether the combination of grass allergen sublingual immunotherapy (SLIT) and dupilumab for 2 years is more effective than double placebo in suppressing the nasal allergen challenge (NAC) response to grass pollen at 1 year after completion of study medication.

DETAILED DESCRIPTION:
This is a double-blind (masked) placebo-controlled trial in adults (N=108 subjects will be enrolled) with moderate to severe seasonal allergic rhinitis and allergic sensitization to grass pollen. Eligible participants who demonstrate a positive response defined by a Total Nasal Symptom Score [TNSS] ≥ 5 (Scale 0-12 in response to a Nasal Allergen Challenge [NAC] with grass pollen extract), will be randomized to one of the following 3 groups in a 1:1:1 ratio:

* Grass allergen sublingual immunotherapy (SLIT) + dupilumab (n=36)
* Grass allergen SLIT +dupilumab placebo (n=36)
* Grass allergen SLIT placebo + dupilumab placebo (n=36)

Grazax® is a sublingual grass allergen immunotherapy product approved for clinical use in the United Kingdom and will be used as SLIT in this study. Grazax (and its matching placebo) will be self-administered daily by participants for a duration of two years.

Dupixent®is the brand name for dupilumab and is a monoclonal antibody against the interleukin 4 (IL-4) receptor. Dupilumab (and its matching placebo) will be administered every two weeks by subcutaneous injection through for a duration of two years, administered by study personnel. The treatment phase of two years will be followed by an observation phase of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to understand and provide informed consent
* A clinical history of grass pollen-induced allergic rhinoconjunctivitis for at least 2 years, with peak symptoms in May, June, or July
* A clinical history of moderate to severe rhinoconjunctivitis symptoms for at least 2 years, interfering with usual daily activities or with sleep as defined according to the Allergic Rhinitis and Its Impact on Asthma (ARIA) classification of rhinitis
* A clinical history of inadequately controlled rhinoconjunctivitis symptoms, despite treatment with antihistamines and/or nasal corticosteroids during the grass pollen season, for at least 2 years
* Positive skin prick test response at screening, defined as wheal diameter ≥3 mm to Phleum pratense
* Positive specific immunoglobulin E (IgE) at screening, defined as IgE class 2 (e.g., ≥ 0.7 kilounits per liter [kU/L]) against Phleum pratense
* A positive response to nasal allergen challenge (NAC) with Phleum pratense defined as a Total Nasal Symptom Score (TNSS) ≥5 points (out of a maximum possibility 12 points)
* A woman of childbearing potential (WOCBP), regardless of birth control history, must:

  * have a negative serum pregnancy test at screening,
  * not be breast-feeding or lactating, and ---is required to consistently use one of the following highly effective methods of contraception throughout the study:

    * hormonal (e.g. oral, transdermal, intravaginal, implant, or injection),
    * intrauterine device (IUD) or system (IUS),
    * vasectomized partner,
    * bilateral tubal occlusion, or
    * sexual abstinence.

Exclusion Criteria:

* Inability or unwillingness of the Subject to give written informed consent or to comply with study protocol requirements
* Prebronchodilator forced expiratory volume (FEV1) <70% of predicted value at either Screening Visit or Baseline (Visit 0) Visit
* A clinical history of asthma requiring regular inhaled corticosteroids for >4 weeks per year, outside of the grass pollen season
* A clinical history of moderate to severe allergic rhinitis, as defined according to the Allergic Rhinitis and Its Impact on Asthma (ARIA) classification of rhinitis, caused by either:

  * An allergen to which the Subject is regularly exposed, or
  * Tree pollen during tree pollen season, treated with regular antihistamine or intranasal corticosteroids
* History of emergency visit or hospital admission for asthma in the previous 12 months
* History of chronic obstructive pulmonary disease
* History of recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment
* History of chronic sinusitis, defined as a sinus symptoms lasting greater than 12 weeks, that includes 2 or more major factors or 1 major factor and 2 minor factors.

  * Major factors are defined as:

    * Facial pain or pressure,
    * Nasal obstruction or blockage,
    * Nasal discharge or purulence or discolored postnasal discharge,
    * Purulence in nasal cavity, or
    * Impaired or loss of smell.
  * Minor factors are defined as:

    * Headache,
    * Fever,
    * Halitosis,
    * Fatigue,
    * Dental pain,
    * Cough, and/or
    * Ear pain, pressure, or fullness.
* History of systemic disease affecting the immune system, such as autoimmune diseases, immune complex disease or immunodeficiency
* At randomization: Current symptoms of, or treatment for:

  * Upper respiratory tract infection,
  * Acute sinusitis,
  * Acute otitis media, or
  * Other relevant infectious process ---Note: 1.) Serous otitis media is not an exclusion criterion and 2.) Participants may be re-evaluated for eligibility after symptoms resolve.
* A past history of any malignant disease in the previous 5 years
* Any tobacco smoking within the last 6 months, or a history of greater than or equal to 10 pack years of cigarette use.
* Any vaping or electronic cigarette use within the last 6 months
* Previous immunotherapy with grass pollen allergen within the previous 5 years
* Previous treatment by dupilumab (Dupixent®)
* Previous Grade 4 anaphylaxis (World Allergy Organization grading criteria), due to any cause
* History of anti-IgE, anti-IL-5, anti-IL-5 receptor, anti-IL-4/IL-13 receptor, or other monoclonal antibody treatment
* Use of tricyclic antidepressants or monoamine oxidase inhibitors
* Ongoing systemic immunosuppressive treatment
* History of intolerance to the study therapy, rescue medications, or their excipients
* For women of childbearing age a positive serum or urine pregnancy test with sensitivity of less than 50 milli-international units per milliliter [mIU/ml] within 72 hours before the scheduled start of study therapy
* The use of any investigational drug within 30 days of the Screening Visit
* The presence of any medical condition that the investigator deems incompatible with participation in the trial
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or may impact the quality or interpretation of the data obtained from the study
* Eosinophilic esophagitis or a diagnosis of any hypereosinophilic syndrome, and/or
* Administration of live attenuated vaccines within four weeks of dupilumab or dupilumab placebo injections, before the first injection and throughout the treatment period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
TNSS Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour After the Challenge (0-1 Hour (hr) at Year 3 | 0 to 1 hour of the NAC at Year 3 (One Year After Completion of Treatment)
  NAC (TNSS Area-under-Curve [AUC 0-1hr]), comparing the TNSS AUC 0-1 hr between the referenced treatment arms: a clinical tolerance outcome measure at Year 3, one year after completion of treatment.
  The Total Nasal Symptom Score (TNSS) is a participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing), each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score is calculated as the sum of the response for all 4 individual nasal symptom scores and can range from a minimum score of 0 to a maximum score of 12: a higher score indicates more severe symptoms.
  The primary treatment comparison is between SLIT/Dupilumab and Double-Placebo.

SECONDARY OUTCOMES:
TNSS Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour After the Challenge (0-1 Hour (hr) at Years 1 and 2 | 0 to 1 hour of the NAC at Years 1 and 2
  NAC (TNSS Area-under-Curve [AUC 0-1hr]), comparing the referenced treatment arms at years 1 and 2 while on study treatment for clinical desensitization.
  The Total Nasal Symptom Score (TNSS) is a participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing), each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score is calculated as the sum of the response for all 4 individual nasal symptom scores and can range from a minimum score of 0 to a maximum score of 12: a higher score indicates more severe symptoms.
  The following treatment comparisons are of secondary outcome interest:
  * Comparison between SLIT/Dupilumab and Double-Placebo
  * Comparison between SLIT/Dupilumab versus SLIT/Dupilumab Placebo
  Both treatment comparisons are key secondary endpoints at Year 2 and therefore multiplicity adjustments are considered; however, at Year 1 the same comparisons are not adjusted for multiplicity.
Peak Nasal Inspiratory Flow (PNIF) (Delta PNIF Area Under the Curve [AUC] 0-1 hr) at Years 1, 2, and 3 | 0 to 1 hour of the NAC at Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  PNIF is defined as the speed of inspiration of air in Liters per minute when breathing into the lungs through the nose. Lower scores indicate less ability to breathe air into the lungs due to more severe nasal congestion.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however, at Years 1 and 2 the comparisons are not adjusted for multiplicity.
TNSS Peak (Maximum) Value Post Nasal Allergen Challenge (NAC) Over the First Hour After the Challenge (0-1 Hour (hr) at Years 1, 2, and 3 | 0 to 1 hour of the NAC at Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  The NAC Total Nasal Symptom Score (TNSS) is a participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing), each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score is calculated as the sum of the response for all 4 individual nasal symptom scores and can range from a minimum score of 0 to a maximum score of 12: a higher score indicates more severe symptoms.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Size of Early Intradermal Skin Test Response at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  An intradermal skin test will be performed using Timothy grass pollen, with an early phase read-out after 15 minutes (with a +/- 3 minute window). A 10 BU test concentration will be used. The average of left and right arm wheal sizes will be used for analysis. A higher wheal size indicates a more severe reaction.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Size of Late Intradermal Skin Test Response at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  An intradermal skin test will be performed using Timothy grass pollen, with a late phase read-out after 6.5 hours (with a +/- 30 minute window) post initial injection. A 10 BU test concentration will be used. The average of left and right arm wheal sizes will be used for analysis. A higher wheal size indicates a more severe reaction.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however, at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Size of Skin Prick Test Endpoint Titration Response as defined by the Provocative Concentration at 5mm (PC5) at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  A skin prick test endpoint titration response assessment will be performed using increasing concentrations of Timothy grass pollen, including: 10 SQ-U/mL, 100 SQ-U/mL, 1000 SQ-U/mL, 10000 SQ-U/mL, and 100000 SQ-U/mL. The average of left and right arm wheal sizes will be used for analysis. The PC5 is defined as the minimum concentration (on the base-10 log scale) for which an average wheal size of 5mm is met or exceeded, based on linear interpolation. A smaller PC5 indicates a more severe reaction.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however, at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Weekly Seasonal Combined Symptom Medication Score (CSMS) at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  A participant-reported seasonal symptoms outcome calculated as an average of: a) weekly Visual Analogue Scale (VAS) score and b) weekly medication score (WMS), each assessed for the 7 days prior to the assessment. The VAS is on a Likert scale (0 to 10 cm, 0=No Symptoms, 10=Worst possible symptoms), reflecting the impact of rhinitis ("hay fever") symptoms. The WMS is based on use of antihistamines (oral and/or eyedrop) and intranasal corticosteroids (score 0 to 10, 0 = medications not used this week, 10 = medications on 5 or more days this week).
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  This treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Weekly Seasonal Visual Analogue Scale (VAS) 0-10 cms Score at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  A participant-reported (self-administered) seasonal symptoms outcome measure on a Likert scale (0 to 10 cm, 0=No Symptoms, 10=Worst possible symptoms), a quality of life measure reflecting the impact of rhinitis ("hay fever") symptoms experienced during the 7 days prior to the assessment.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, no comparisons at any year are adjusted for multiplicity for this outcome.
Weekly Seasonal Medication Score (WMS) at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  A participant-reported (self-administered) seasonal symptoms medications score based on the use of antihistamines (oral and/or eyedrop) and intranasal corticosteroids, assessed for the 7 days prior to the assessment. The WMS has a score ranging from 0 to 10 (0 = medications not used this week, 10 = medications on 5 or more days this week).
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, no comparisons at any year are adjusted for multiplicity for this outcome.
Weekly Rhinitis Quality of Life Score Using the Juniper Mini-Rhinoconjunctivitis Quality of Life Questionnaire (miniRQLQ) at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  The Juniper Mini-Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ), is a participant-reported (self-administered) questionnaire that consists of 14 questions grouped into 5 domains. Each question is scored on a scale of 0 (not troubled with symptoms) to 6 (extremely troubled with symptoms) and describes nose/eye symptoms experienced for the 7 days prior to the assessment. A total score equal to the average of all questions will be analyzed.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Modified Rhinitis Symptom Utility Index (MRSUI) Questionnaire Measured In-Season at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  The Modified Rhinitis Symptom Utility Index (MRSUI) questionnaire consists of 10 questions regarding symptoms experienced during the prior 2 weeks from the nose, eyes, and throat, specifically how frequently the symptoms occurred and how bothersome they were. The total MRSUI score will be calculated as the sum of the numeric responses to all 10 questions. Higher scores indicate a worse outcome, where the maximum score is 25.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Global Evaluation Questionnaire Number 1 at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  Participants are asked to describe their allergic rhinitis ("hay fever"). This administered questionnaire is comprised of 6 questions, focusing on nasal and eye symptoms [0=No symptoms, 3=Severe]. The total Global Evaluation No. 1 score will be calculated as the total sum of the numeric responses to all 6 questions. Higher scores indicate a worse outcome/severity, where the maximum score per visit is 18.
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however, at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Global Evaluation Questionnaire Number 2 at Years 1, 2, and 3 | Years 1 and Year 2, and at Year 3 (One Year After Completion of Treatment)
  For the Global Evaluation No. 2 questionnaire, participants are asked a single question regarding the change in current rhinitis/hay fever compared to the years prior to initiating study treatment (Much better: +3, Much worse: -3).
  The following treatment comparison is of secondary outcome interest, where Year 3 is a clinical tolerance outcome measure, and Years 1 and 2 are clinical desensitization outcome measures:
  • Comparison between SLIT/Dupilumab and Double-Placebo
  According to the SAP, this treatment comparison at Year 3 is a key secondary endpoint and therefore a multiplicity adjustment is considered; however at Years 1 and 2 the comparisons are not adjusted for multiplicity.
Frequency, Severity, and Relatedness of Treatment-Emergent Adverse Events (AEs) by Treatment Arm | Start of study treatment until completion of study participation at year 3, or until 30 days after prematurely withdrawing from the study
  The number and percentage of participants with at least one treatment-emergent AE in the following categories will be summarized by treatment arm:
  1. any AE related to any study drug
  2. any severe (Grade 3 or higher) AE
  Only treatment-emergent AEs will be summarized. All AEs, including local, systemic, and serious AEs will be considered. For grading severity, the protocol-specified grading criteria will be used which depends on the type of AE:
  * Grading Table for Local Reactions to SLIT (Grades 1-4)
  * Grading Table for Local Reactions to Allergen Skin Testing (Grades 1-3)
  * Grading Table for NAC Procedure for Local Reactions (Grades 1-4)
  * WAO Subcutaneous Immunotherapy Systemic Reaction Grading System (Grades 1-5) for any immediate (0-1hr) systemic allergic reaction
  * National Cancer Institute's (NCI's) Common Toxicity Criteria for Adverse Events (CTCAE) v5.0 (November 27, 2017; Grades 1-5) for all remaining AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Durham, MD, Study Chair — Allergy and Clinical Immunology Section at NHLI,Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org

DOCUMENTS (1):
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04502966/ICF_000.pdf